CLINICAL TRIAL: NCT02816125
Title: Effects of Omega-3 Fatty Acids on Risk Factors for Breast Cancer in Pre-menopausal Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Guelph (Other)
Collaborators: Alison Duncan (Unknown)
Responsible Party: Principal Investigator, Kelly Anne Meckling, PhD, Professor, University of Guelph
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 235
Record Dates: First submitted 2016-06-24; First posted 2016-06-28 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Healthy; Premenopausal Period
Keywords: breast cancer; fatty acids; omega-3
MeSH Terms: conditions — Breast Neoplasms | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Habitual supplemented (Active Comparator): habitual diet with 1.2 g EPA+DHA in capsule form/day.
  Interventions: Dietary Supplement: omega-3 fatty acid
- Low-fat supplemented (Experimental): Reduce dietary fat to less than 20% energy, add 1.2 g EPA+DHA in capsule form/day.
  Interventions: Dietary Supplement: omega-3 fatty acid

INTERVENTIONS:
Dietary Supplement: omega-3 fatty acid — SEE YOURSELF WELLTM OMEGA-3 Dietary Supplement: See Yourself Well Inc., Leamington, Ontario) containinged 200 mg of EPA and 100 mg of DHA for a total of 1.2 g n-3/day.

SUMMARY:
Healthy premenopausal women were enrolled in a diet intervention study that examined the effect of a combination EPA/DHA supplement on risk factors associated with breast cancer. In a randomized cross-over design, women consumed their habitual diet with a supplement for three menstrual cycles, had three cycles of wash-out and then consumed a low-fat diet with the same supplement. Blood, urine and nipple aspirate fluid were collected periodically over the 10 month protocol and analyzed for biomarkers associated with supplementation and future risk of breast cancer.

DETAILED DESCRIPTION:
Non-pregnant, non-lactating women aged 18+ were recruited by way of posters, to take part in a dietary intervention study that was examining the effects of dietary fat level and fat type on risk factors associated with breast cancer. Women who were normally menstruating, consumed either their habitual diet or a low-fat diet for three menstrual cycles, along with a supplement containing 1.2 g DHA+EPA /day. This was followed by a 3-menstrual cycle washout, where the habitual diet was consumed without a supplement. Subsequently the participants consumed the other diet (either low-fat or habitual) for a further 3 menstrual cycles with the 1.2 g DHA/EPA supplement. Blood, urine and nipple aspirate fluid were collected at the beginning and end of each intervention period and analyzed for a variety of biomarkers. Diet records were collected continuously over the entire study period and periodic 7-day records examined for collection of detailed nutrition information. Anthropometry was completed at each study visit, and nutritional counselling provided throughout.

ELIGIBILITY:
Inclusion Criteria: menstruating, pre-menopausal -

Exclusion Criteria: pregnant, lactating, post-menopausal, smoking, on birth control pills

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2004-03; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
omega-3 fatty acid incorporation into red blood cells | 3 months
  replacement of omega-6 long chain fatty acids with DHA and EPA in red blood cell membranes
omega-3 fatty acid incorporation in cell material from nipple aspirate fluid | 3 months
  replacement of omega-6 fatty acids with omega-3 fatty acids in the cells sloughed into the ductal fluid and collected. Total fatty acids from PL fraction of NAF.

SECONDARY OUTCOMES:
changes in estrogen in blood and nipple aspirate fluid | 3 months
  modification of estrogen production following omega-3 fatty acid consumption
changes in oxidative estrogen metabolites in urine | 3 months
  lower concentrations of oxidized estrogen metabolites expected with omega-3 fatty acid supplementation.
Body weight changes | 1 month
  lower body weight expected with implementation of the low-fat diet

CONTACTS AND LOCATIONS:
Overall Officials: Sandy Auld, MSc, Study Director — Research Ethics Officer, University of Guelph

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gomes MA, Jia X, Kolenski I, Duncan AM, Meckling KA. The role of background diet on the effects of eicosapentaenoic acid and docosahexaenoic acid supplementation in healthy pre-menopausal women: a randomized, cross-over, controlled study. Lipids Health Dis. 2016 Sep 29;15(1):168. doi: 10.1186/s12944-016-0341-1. PMID 27687127